CLINICAL TRIAL: NCT03222271
Title: Intelligent Volume Assured Pressure Support (iVAPS) vs. Spontaneous/Timed Mode as Noninvasive Modes for Weaning of COPD Patients
Brief Title: iVAPS vs. S/T Modes as Non-invasive Weaning Strategy in COPD Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Sarah Mohammed Hashem Hamza Ahmed, Pricipal Investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IVAPSSTMNMWCP
Record Dates: First submitted 2017-07-13; First posted 2017-07-19 (Actual); Last update posted 2021-01-13 (Actual); Status verified 2021-01

CONDITIONS: COPD Exacerbation
Keywords: NIV weaning strategy

STUDY DESIGN:
Intervention Model Description: All patients will be subjected to history and clinical examination,severity assessment(mMRC dyspnea scale,APACHE II Score and CAT score).
  A) Extubation to NIV: SBT will be attempted once the patients achieve stability regarding clinical, neurological and biochemical parameters.Failure of SBT is considered if:pH < 7.35,PaCO2 > 15-20% increase above baseline,PaO2 < 50 mmHg.Heart rate > 100 bpm or respiratory rate > 35 cycle/min.
  * RSBI and P 0.1. will be recorded while on SBT
  B) The patients will be randomized to receive NIV using either ST or iVAPS mode.
  C) The patients will be categorized in analysis into 3 groups,Group I: Simple weaning ,Group II: Difficult weaning and Group III: Prolonged weaning.
  -The following parameters will be recorded for the patients at the beginning of the study and at 1, 2, 12, 24 and 48 hours after initiation of NIV therapy:GCS,Vital signs (HR, SBP& DBP,RR), ABG analysis and Patient's comfort.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- I) Extubation to NIV (S/T mode) (Active Comparator): The patients will receive NIV using S/T mode after extubation with the following parameters:
  * Expiratory Positive Airway Pressure (EPAP): 4-8 centimeter water (cmH2O).
  * Inspiratory Positive Airway Pressure (IPAP): 12-20 cmH2O.
  * Respiratory rate (RR): 10-12 breath/minute.
  Interventions: Device: Extubation to NIV
- II) Extubation to NIV (iVAPS) mode (Experimental): The patients will receive NIV using iVAPS mode after extubation with the following parameters:
  * Patient's height in cm..
  * Target alveolar ventilation (Va): adjusted provided that tidal volume is 8 ml/kg of ideal body weight (IBW).
  * Expiratory Positive Airway Pressure (EPAP) :4-8 cmH2O
  * Minimum and maximum Pressure Support (PS) :8-16
  * Respiratory rate :10-12 breath/min.
  Interventions: Device: Extubation to NIV

INTERVENTIONS:
Device: Extubation to NIV — Weaning using NIV immediately after extubation with the mentioned parameters
  Other Names: NIV portable device: Res MED(S9 VPAPTM ST)

SUMMARY:
Invasive mechanical ventilation (IMV) is associated with numerous complications. Hence, patients should be weaned from the ventilator as early as possible. A number of randomized controlled trials have addressed whether noninvasive ventilation (NIV) can facilitate weaning in patients failing spontaneous breathing trials (SBT)s. Compared to invasive weaning, NIV weaning strategy showed reduced mortality, greater weaning success, less ventilator-associated pneumonia, shorter length of ICU and hospital stay and less re-intubation rate.

Most of the previous studies used pressure support ventilation with fixed pressure support, but no studies published on hybrid NIV modes.

Intelligent Volume Assured Pressure Support (iVAPS) is a recent NIV mode, which achieves a target alveolar ventilation by adjusting pressure support and respiratory rate automatically. In iVAPS, the target is alveolar ventilation not the tidal volume, taking into account a predicted dead space . This new mode has been investigated in stable chronic obstructive pulmonary disease (COPD) patients with domiciliary NIV and it was comparable to pressure support ventilation (PSV) regarding improvement in oxygenation, carbon dioxide (CO2) wash and therapy compliance.

Yet, less numerous studies have been performed on this mode when used for acute respiratory failure. These studies found that i-VAPS was comparable to PSV as regards PaCO2 and pH improvements, minute volume, pressure support and respiratory rate. No published data so far about the role of i-VAPS as a weaning mode in mechanically ventilated patients. So, this study aims to investigate this new mode in comparison to the standard S/T mode in weaning COPD patients using NIV.

DETAILED DESCRIPTION:
Invasive mechanical ventilation (IMV) is associated with numerous complications. Hence, patients should be weaned from the ventilator as early as possible . Approximately 25% and (14-22) % of mechanically ventilated patients experience difficult and prolonged weaning respectively. A number of randomized controlled trials have addressed whether NIV can facilitate weaning in patients failing SBTs. The most recent systemic review included 16 trials -mainly COPD patients- found that patients weaned with NIV had reduced mortality, greater weaning success, less ventilator-associated pneumonia, shorter length of ICU and hospital stay and less reintubation rate.

Most of the previous studies used pressure support ventilation with fixed pressure support, but no studies published on hybrid NIV modes. Intelligent Volume Assured Pressure Support (iVAPS) is a recent NIV mode, which achieves a target alveolar volume by adjusting pressure and respiratory rate automatically. In iVAPS, the target is alveolar ventilation not the tidal volume. taking into account a predicted dead space. This new mode has been investigated in stable COPD patients with domiciliary NIV and it was comparable to pressure support ventilation (PSV) regarding improvement in oxygenation, CO2 wash and therapy compliance. Other studies focused on sleep quality and found that iVAPS was comparable to PSV regarding sleep quality, arousal, O2 de-saturation index, increase in therapy adherence and decrease in median PS needed with iVAPS.

Yet, less numerous studies have been performed on this mode when used for acute respiratory failure. These studies investigated the outcomes in acute hypercapnic respiratory failure and found that iVAPS was comparable to PSV as regards PaCO2 and logarithm of hydrogen ion concentration (pH) improvements, minute volume, pressure support and respiratory rate. No published data about the role of iVAPS as a weaning mode in mechanically ventilated patients.

ELIGIBILITY:
Inclusion Criteria:

All patients in acute exacerbation of COPD who are mechanically ventilated will be included in this study.

Exclusion Criteria:

* Age < 18 years or >75 years.
* Other chest diseases (pneumonia, bronchiectasis, pulmonary embolism, pulmonary fibrosis…).
* Tracheostomized patients.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2017-10-25 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2020-09-30 (Actual)

PRIMARY OUTCOMES:
Success rate of either modes. | 48 hours
  -Success is considered when the patient is able to achieve the following: pH >7.35,decrease in partial pressure of carbon dioxide (PaCO2) of >15-20%, partial pressure of oxygen (PaO2)>60 mmHg, arterial oxygen saturation (SaO2)> 90% on fraction of inspired oxygen (FiO2) <40%, RR < 24 bpm and no signs of respiratory distress like agitation, diaphoresis or anxiety.
  Numbers of successful cases is recorded

SECONDARY OUTCOMES:
Re-intubation rate in each group. | 30 days
  Measured by number of the patients re-intubated in each arm
Mortality rate in each group | 30 days
  Measured by number of the patients re-intubated in each arm
Duration spent on NIV | An average of 30 days
  Measured in days
Length of ICU stay | An average of 30 days
  Measured in days
Degree of patient's comfort | An average of 30 days
  A specific questionnaire (pain in the forehead, nose, cheeks, and chin, air leak at eyes and mouth, dry nose and mouth, skin inflammation and claustrophobia. The patients answers to each question (sore0-3 in terms of intensity). The total score is calculated by adding the individual scores of each item mentioned above.

CONTACTS AND LOCATIONS:
Overall Officials: Suzan S Sayed, MD, Study Chair — Assiut University; Aliaë A. Mohamed-Hussein, MD, Study Director — Assiut University; Doaa M Magdy, MD, Study Director — Assiut University; Sarah M Hamza, MSc, Principal Investigator — Assiut University
Locations (2):
- Egypt (2):
  - Assiut University Hospital, Asyut
  - Assiut University Hospital - RICU, Asyut

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Funk GC, Anders S, Breyer MK, Burghuber OC, Edelmann G, Heindl W, Hinterholzer G, Kohansal R, Schuster R, Schwarzmaier-D'Assie A, Valentin A, Hartl S. Incidence and outcome of weaning from mechanical ventilation according to new categories. Eur Respir J. 2010 Jan;35(1):88-94. doi: 10.1183/09031936.00056909. Epub 2009 Jun 18. PMID 19541716
- [Background] Burns KE, Meade MO, Premji A, Adhikari NK. Noninvasive ventilation as a weaning strategy for mechanical ventilation in adults with respiratory failure: a Cochrane systematic review. CMAJ. 2014 Feb 18;186(3):E112-22. doi: 10.1503/cmaj.130974. Epub 2013 Dec 9. PMID 24324020
- [Background] Talwar D, Dogra V. Weaning from mechanical ventilation in chronic obstructive pulmonary disease: Keys to success. J Assoc Chest Physicians 2016;4:43-9.
- [Background] Kelly JL, Jaye J, Pickersgill RE, Chatwin M, Morrell MJ, Simonds AK. Randomized trial of 'intelligent' autotitrating ventilation versus standard pressure support non-invasive ventilation: impact on adherence and physiological outcomes. Respirology. 2014 May;19(4):596-603. doi: 10.1111/resp.12269. Epub 2014 Mar 24. PMID 24661390
- [Background] Battisti A, Tassaux D, Bassin D, Jolliet P. Automatic adjustment of noninvasive pressure support with a bilevel home ventilator in patients with acute respiratory failure: a feasibility study. Intensive Care Med. 2007 Apr;33(4):632-8. doi: 10.1007/s00134-007-0550-1. Epub 2007 Feb 24. PMID 17323049